CLINICAL TRIAL: NCT06754371
Title: Safety and Efficacy of Prophylactic Tranexamic Acid in Reducing Postpartum Hemorrhage After Cesarean Delivery in Women with Systemic Autoimmune Disease：A Randomized Controlled Trial
Brief Title: Prophylactic Tranexamic Acid Reduces Postpartum Hemorrhage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LY2024-172-B
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hemorrhage; Systemic Autoimmune Diseases
Keywords: postpartum hemorrhage; systemic autoimmune disease; cesarean delivery; thromboembolism
MeSH Terms: conditions — Postpartum Hemorrhage; Thromboembolism | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid group (Experimental): intravenous infusion of tranexamic acid 1g (20ml) 10min before skin dissection
  Interventions: Drug: tranexamic acid
- Placebo group (Placebo Comparator): intravenous infusion of normal saline 20ml 10min before skin dissection
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: tranexamic acid — intravenous infusion of tranexamic acid 1g (20ml) 10min before skin dissection
  Other Names: TXA
  Arms: Tranexamic acid group
Drug: normal saline — intravenous infusion of normal saline 20ml 10min before skin dissection
  Arms: Placebo group

SUMMARY:
Postpartum hemorrhage (PPH) is the most significant leading cause of pregnancy-related mortality in high-risk cesarean delivery women. Systemic autoimmune diseases are associated with adverse pregnancy outcomes (APOs), including PPH, preeclampsia, thromboembolism, abortion, and intrauterine growth restriction. The incidence of PPH in women with systemic lupus erythematosus has been reported to be as high as 34%. Prevention of PPH is the key to reduce complications in high-risk women. In recent years, a large number of clinical studies have confirmed that the early preventive use of tranexamic acid(TXA) can reduce the amount of blood loss, the need for additional uterine contraction agents, the risk of blood transfusion, and maternal adverse outcomes, and do not increase the risk of thromboembolic events, which can be used to prevent PPH. However, the study population of TXA is mainly low-risk puerpera, and there is still a lack of relevant research on TXA used in pregnant women with systemic autoimmune diseases. The purpose of this study was to evaluate the safety and efficacy of TXA in preventing postpartum hemorrhage after cesarean delivery in women with systemic autoimmune disease, as well as the maternal and neonatal risks associated with systemic autoimmune disease, to provide evidence for clinical practice and further research.

DETAILED DESCRIPTION:
The worldwide estimated cumulative prevalence of autoimmune disease is approximately 5%. Studies are often limited by small sample sizes and focused on a specific autoimmune disease such as systemic lupus erythematosus (SLE) and antiphospholipid syndrome (APS), which is characterized by the production of autoantibodies leading to inflammation of multiple organs. Systemic autoimmune diseases are associated with adverse pregnancy outcomes (APOs), including increased cesarean delivery rates, PPH, preeclampsia, thromboembolism, abortion, premature delivery, and intrauterine growth restriction. Preeclampsia is the most commonly reported complication in patients with SLE and is also a high risk factor for PPH. The incidence of PPH in women with SLE has been reported to be as high as 34%. PPH increases the need for blood transfusion and related complications and is a significant clinical and socio-economic problem. Therefore, prevention of PPH is the key to reduce the postpartum complications of high-risk women. At present, the methods commonly used to prevent PPH after cesarean delivery include uterine massage, prophylactic use of uterine contraction agents in the third stage of labor, and early use of TXA. Recent clinical studies of TXA use in high-risk cesarean delivery women have shown that prophylactic use of TXA significantly reduces blood loss, prevents PPH, and reduces ICU admission and length of stay. There was no evidence of an increased risk of maternal-related complications with TXA use. But there is still a lack of relevant research on TXA used in pregnant women with systemic autoimmune diseases. Anti-phospholipid antibodies (aPL) are often present in SLE and APS patients, which predict serious perinatal complications and are associated with the risk of thrombosis. aPL are detected not only in SLE and APS but also in other connective tissue diseases such as systemic sclerosis (SSc), Sjögren's syndrome (SS), rheumatoid arthritis (RA), and undifferentiated connective tissue disease (UCTD). Although TXA has been widely used in patients at high risk for thromboembolism, such as trauma, orthopedics, and cardiac surgery in recent years, the evidence strongly supports that it does not increase the risk of death or thromboembolic complications. More evidence from high quality randomized controlled trials is needed to assess the benefits and risks of its use in women at high risk of PPH after cesarean delivery.

The aim of this study was to evaluate the safety and efficacy of TXA in preventing PPH after cesarean delivery in women with systemic autoimmune disease. Patients undergoing cesarean delivery were randomly assigned to TXA group(intravenous infusion of TXA 1g (20ml) 10min before skin dissection) and placebo group(intravenous infusion of normal saline 20ml 10min before skin dissection).The estimated blood loss 24h postoperatively, blood transfusion 3d postpartum, additional uterotonics, other surgical intervention for PPH and thromboembolic events were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cesarean delivery
2. Preoperative diagnosis of pregnancy with systemic autoimmune diseases (systemic lupus erythematosus, antiphospholipid syndrome, systemic sclerosis, Sjogren's syndrome, rheumatoid arthritis, undifferentiated connective tissue disease)
3. Obtain informed consent.

Exclusion Criteria:

1. intrauterine fetal death
2. Existing/previous history of thromboembolism
3. Hemorrhagic disease, significant prenatal bleeding
4. Balloon placement of internal iliac artery
5. Allergic to tranexamic acid
6. Severe renal insufficiency (serum creatinine >451μmol/L or blood urea nitrogen >20mmol/L)
7. Epilepsy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of postpartum hemorrhage | From skin incision to 1day after surgery
  Postpartum hemorrhage is defined as blood loss of 1000 mL or more within the first 24 h after cesarean delivery.
Estimated blood loss within 1day after surgery | From skin incision to 1day after surgery
  Estimated blood loss is calculated by GROSS EQUATION: Estimated Blood Loss (EBL) = EBV ×((HCT1 - HCT2)/(HCT mean)), EBV = Estimated Blood volume; whereas EBV = Patient's weight (in kilogram) × 70 mL/kg, HCT1=preoperative hematocrit, HCT2 = postoperative hematocrit, and HCT mean = (HCT1 + HCT2)/2;

SECONDARY OUTCOMES:
The volume of blood transfusion within 3days after surgery and complications | From skin incision to 3days after surgery
  The volume of blood transfusion within 3days after surgery and complications(such as fever, allergy, hemolysis, renal dysfunction，etc）
Whether additional uterotonics are needed | From the delivery of placenta until 3 days postoperatively
  Uterotonics other than intraoperative routine dose intravenous and intrauterine infusion of oxytocin.
Whether other surgical intervention for PPH are needed | From the delivery of placenta until 3 days postoperatively
  Patients who need other surgical intervention(such as intrauterine balloon compression hemostasis, uterine artery ligation or embolization and hysterectomy) to control PPH
Incidence of thromboembolic events | Patients will be followed up to one week after surgery
  The occurrence of thromboembolic events within one week of delivery, including deep vein thrombosis, pulmonary embolism, myocardial infarction, and stroke
Maternal complications | Patients will be followed up to 3days after surgery
  Occurrence of adverse effects (nausea, vomiting, headache, epilepsy, renal impairment，coagulopathy) within 3days after surgery.
Maternal and neonatal 3 months mortality | Patients and neonates will be followed up to 3 months after surgery
  All-cause 3 months mortality
Estimated intraoperative blood loss | From skin incision to the end of the surgery
  Estimated intraoperative blood loss is calculated using the formula: collected blood volume in the suction canister (ml)-the volume of amniotic fluid (ml)-the volume of flushing (ml) + the volume from the gauze tampon (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Xiao, PHD, Study Director — Renji Hospital, Shanghai Jiaotong University, School of Medcine
Locations (1):
- Renji Hospital, Shanghai Jiaotong University, School of Medcine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No